CLINICAL TRIAL: NCT03040947
Title: MRI Sequence and Imaging Protocol Development
Acronym: BikeMRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/2050
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2020-06

CONDITIONS: Cardiomyopathy, Hypertrophic; Cardiomyopathy, Dilated; Left Ventricular Hypertrophy; Ischemic Heart Disease; Hypertension
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Cardiomyopathy, Dilated; Hypertrophy, Left Ventricular; Myocardial Ischemia; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected from all participants before and after the CMR scan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteer: Healthy Volunteers will undergo a cardiovascular magnetic resonance imaging scan.
  Interventions: Other: Cardiovascular Magnetic Resonance
- Diseased (Suspected or Known Cardiac Conditions): Patients will undergo a cardiovascular magnetic resonance imaging scan.
  Interventions: Other: Cardiovascular Magnetic Resonance

INTERVENTIONS:
Other: Cardiovascular Magnetic Resonance

SUMMARY:
The purpose of this study is to develop imaging protocols when using cardiovascular magnetic resonance (CMR) to assess cardiac functions, morphology and tissue characterization. The National Heart Research Institute Singapore (NHRIS) houses two dedicated CMR scanners to support the numerous investigator initiated projects in patients with various cardiac pathologists. By optimizing novel CMR sequences used in these studies, scanning time can be shortened for patients with underlying cardiac diseases.

DETAILED DESCRIPTION:
In medical research, there is a continuous need to develop new imaging techniques such as cardiovascular magnetic resonance (CMR) imaging. This will allow us to visualize and study the function and structure of the heart in greater detail so as to improve the diagnosis and treatment of patients with various cardiac conditions. The aim of the study is to optimise new CMR sequences, allowing the development of imaging protocols in future research studies.

This study will hence recruit 800 subjects for each of the following sub-studies:

1. Sub-study 1: Normal CMR protocols for assessment of cardiac function and morphology
2. Sub-study 2: Exercise stress protocols with a CMR-compatible supine bike.

For the first sub-study, 400 healthy volunteers and patients with cardiac conditions or suspected to have cardiac conditions will be recruited. The testing and optimising of CMR sequence settings are crucial to ensure the accuracy and robustness of the scan before using the scan as a clinical diagnostic tool.

For the second sub-study, 400 healthy volunteers of different fitness levels and and patients with cardiac conditions or suspected to have cardiac conditions will be recruited. An exercise stress protocol will then be developed for future studies in patients with suspected coronary artery diseases. For this protocol, participants will be asked to cycle on a supine exercise bike to assess the effects of exercise and free breathing on the stability of the CMR imaging sequences.

ELIGIBILITY:
Inclusion Criteria:

* Has no known significant medical history
* Is able to give informed consent

Exclusion Criteria:

* Has contraindications to CMR implantable devices, cerebral aneutysm clips and cochlear implants
* Has claustrophobia
* Females who are pregnant
* Is unable to comply with study protocols

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential participants will be identified from an existing database of healthy volunteers who had previously participated in the biobank program and indicated interest in future studies.
  Potential patients are identified from the imaging or admissions databases. The primary physicians of these patients identified will be notified prior to recruitment and the patient will only be recruited if the primary physician is agreeable.
  Alternatively, other methods of participant identification include co-workers of the department who volunteer themselves and indicate on the Informed Consent Document that their participation was entirely voluntary and not under coercion.
  Team members of this study are not eligible for participation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-03; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
First occurrence of cardiovascular event | 1 day
  This outcomes are obtained via hospital records or by a phone follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Le TT, Bryant JA, Ting AE, Ho PY, Su B, Teo RC, Gan JS, Chung YC, O'Regan DP, Cook SA, Chin CW. Assessing exercise cardiac reserve using real-time cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2017 Jan 23;19(1):7. doi: 10.1186/s12968-017-0322-1. PMID 28110638